CLINICAL TRIAL: NCT01714817
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of BMS-188667 (Abatacept) or Placebo on a Background of Mycophenolate Mofetil and Corticosteroids in the Treatment of Subjects With Active Class III or IV Lupus Nephritis
Brief Title: Efficacy and Safety Study of Abatacept to Treat Lupus Nephritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to meet protocol objectives.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-291; 2012-000714-11 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Abatacept; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMS-188667 + Mycophenolate mofetil + Prednisone (Experimental): BMS-188667 30 mg/kg injection by intravenous on Days 1,15, 29, and 57, followed by a weight-tiered dose approximating 10mg/kg injection by intravenous every 4 weeks, Mycophenolate mofetil 1.5 g tablet by mouth and Prednisone up to 60 mg tablet by mouth Daily for 104 weeks
  Interventions: Biological: BMS-188667; Drug: Mycophenolate mofetil; Drug: Prednisone
- Placebo + Mycophenolate mofetil + Prednisone (Placebo Comparator): Placebo matching with BMS-188667 injection by intravenous on Days 1,15, 29, and 57, followed by every 4 weeks, Mycophenolate mofetil 1.5 g tablet by mouth and Prednisone up to 60 mg tablet by mouth Daily for 104 Weeks
  Interventions: Drug: Mycophenolate mofetil; Drug: Prednisone; Biological: Placebo matching with BMS-188667

INTERVENTIONS:
Biological: BMS-188667
  Other Names: Abatacept
  Arms: BMS-188667 + Mycophenolate mofetil + Prednisone
Drug: Mycophenolate mofetil
  Other Names: Cellcept
Drug: Prednisone
Biological: Placebo matching with BMS-188667
  Arms: Placebo + Mycophenolate mofetil + Prednisone

SUMMARY:
The purpose of this study is to evaluate (Abatacept) for treatment of lupus nephritis when used on a background of Cellcept (mycophenolate) and prednisone (corticosteroids)

ELIGIBILITY:
For additional information please contact the BMS Lupus Nephritis Clinical Trial Matching Service at 855-56-LUPUS. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Note: Subjects > 16 are eligible for enrollment at selected centers

Inclusion Criteria:

* Potential subjects must have active lupus nephritis
* Biopsy within 12 months prior to screening visit indicating active Class 3 or 4 proliferative lupus glomerulonephritis (lupus effecting your kidney)
* Urine protein creatinine ratio (UPCR) ≥ 1 at Screening
* Serum creatinine ≤ 3 mg/dL (ie, ≤ 265 micromol/L)
* There must also be evidence of active disease within 3 months of Screening, based on at least one of the following:

  * Worsening of lupus nephritis OR
  * UPCR ≥ 3 at Screening OR
  * Active urine sediment OR
  * Biopsy within 3 months prior to screening visit indicating active Class 3 or Class 4 active proliferative lupus glomerulonephritis

Inclusion Criteria for the Long-Term Extension Period:

* Signed Written Informed Consent
* Subjects who achieve a complete or partial renal response after completing 2 years of double-blind treatment

Exclusion Criteria:

* Systemic Lupus Erythematosus (SLE) must be the primary/main autoimmune diagnosis
* Current symptoms of severe, progressive, or uncontrolled non-SLE related renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological, or cerebral disease, or other concomitant medical conditions that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study
* Significant active Central nervous system (CNS) lupus with the exception of fatigue or mild stable cognitive
* Subjects who are diagnosed as end-stage renal disease or whose kidney damage is too significant and irreversible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (136):
- United States (26):
  - University Of Alabama At Birmingham (Uab), Birmingham, Alabama
  - Valerius Med Group & Res Ctr Of Greater Long Beach, Inc., Long Beach, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - University Of Connecticut Health Center, Farmington, Connecticut
  - University Of Miami Miller School Of Medicine, Miami, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Emory University., Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Tulane University School Of Medicine, New Orleans, Louisiana
  - Brigham & Women'S Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Local Institution, Camden, New Jersey
  - Suny Downstate Medical Center, Brooklyn, New York
  - Northshore Lij Health System, Great Neck, New York
  - The Feinstein Institute For Medical Research, Manhasset, New York
  - Hospital For Special Surgery, New York, New York
  - Local Institution, New York, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Shanahan Rheum & Immunotherapy, PLLC, Raleigh, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - Rheumatology Consultants Pllc, Knoxville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University Of Utah Hospital, Salt Lake City, Utah
  - Local Institution, Charlottesville, Virginia
- Argentina (4):
  - Organizacion Medica De Investigacion S.A. (Omi), Capital Federal, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Buenos Aires
  - Hospital Privado-Centro Medico De Cordoba S.A., Córdoba
- Australia (3):
  - Local Institution, Adelaide, South Australia
  - Local Institution, Parkville, Victoria
  - Local Institution, Perth, Western Australia
- Brazil (7):
  - Local Institution, Savaldor, Estado de Bahia
  - Local Institution, Goiânia, Goiás
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Uberlândia, Minas Gerais
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo
- Canada (2):
  - Local Institution, Mississauga, Ontario
  - Local Institution, Toronto, Ontario
- Chile (3):
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Independencia, Santiago Metropolitan
  - Local Institution, Santiago, Santiago Metropolitan
- China (19):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Haikou, Hainan
  - Local Institution, Wuhan, Hebei
  - Local Institution, Harbin, Heilongjiang
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Wuxi, Jiangsu
  - Local Institution, Nanchang, Jiangxi
  - Local Institution, Xi'an, Shan1xi
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Beijing
  - Local Institution, Chongqing
  - Local Institution, Guangzhou
  - Local Institution, Nanchang
  - Local Institution, Nanning
  - Local Institution, Shanghai
  - Local Institution, Xi'an
- Colombia (6):
  - Riesgo De Fractura S.A. Cayre Ips, Bogota, Cundinamarca
  - Servimed E.U, Bucaramanga, Santander Department
  - Clinica De La Costa, Barranquilla
  - Circaribe S.A.S, Barranquilla
  - Hospital Universitario San Ignacio, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
- Local Institution, Prague, Czechia
- Local Institution, Hong Kong, Hong Kong
- India (6):
  - Local Institution, Secunderabad, Andhra Pradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Gūrgaon
  - Local Institution, Hyderabad
  - Local Institution, Lucknow
  - Local Institution, New Delhi
- Israel (3):
  - Local Institution, Haifa
  - Local Institution, Ramat Gan
  - Local Institution, Tel Aviv
- Italy (5):
  - Local Institution, Brescia
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Reggio Emilia
  - Local Institution, Torino
- Japan (22):
  - Local Institution, Nagakute-shi, Aichi-ken
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Chiba, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Maebashi, Gunma
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Sendai, Miyagi
  - Local Institution, Nagasaki, Nagasaki
  - Local Institution, Niigata, Niigata
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Shimotsuke-shi, Tochigi
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Fuchū, Tokyo
  - Local Institution, Ōta-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Kita-gun
  - Local Institution, Osaka
- Mexico (9):
  - Local Institution, Mexico City, Distrito Fededral
  - Centro De Est D Inv. Basica Y Clinica, Guadalajara, Jalisco
  - Local Institution, Guadalajara, Jalisco, Jalisco
  - Hospital De Jesus, Mexico City, Mexico City
  - Hospital General De Mexico O.D., Mexico City, Mexico City
  - Centro Medico De Las Americas, Mérida, Yucatán
  - Instituto Nacional De Ciencias Medicas Y Nutricion S.Z., Distrito Federal
  - Centro Potosino de Inv Clinica, San Luis Potosí City
  - Hosp Central I.Morones Prieto, San Luis Potosí City
- Peru (3):
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - Instituto De Ginecologia Y Reproduccion Inv. Clinical Sac, Lima
- Local Institution, San Juan, Puerto Rico
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
  - Local Institution, Iași
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Ufa
- South Korea (2):
  - Local Institution, Daegu
  - Local Institution, Seoul
- Local Institution, Madrid, Spain
- Taiwan (4):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Turkey (Türkiye) (2):
  - Local Institution, Antalya
  - Local Institution, Edirne

REFERENCES:
- [Derived] O'Connor SK, Devarajan P, Liu J, Maldonado MA, Sproles A, Rose J, Thornton S, Chen C, Huang B, Brunner HI. The Renal Activity Index for Lupus: Validation for Prediction of Kidney Inflammation in Adult Patients With Lupus Nephritis. J Rheumatol. 2026 Jan 15:jrheum.2025-0504. doi: 10.3899/jrheum.2025-0504. Online ahead of print. PMID 41241398
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 695 participants were enrolled; 406 randomized; and 405 received treatment. 289 participants were screen failures and never treated with study medication; 233 were due to no longer meeting study criteria; 19 withdrew consent; 4 due to Adverse Events; 1 due to death; 1 due to poor/non-compliance; 1 was lost to follow up; and 30 were other.
Groups:
- Abatacept IV: Abatacept 30 mg/kg injection by intravenous on Days 1,15, 29, and 57, followed by a weight-tiered dose approximating 10mg/kg injection by intravenous every 4 weeks, Mycophenolate mofetil 1.5 g tablet by mouth and Prednisone up to 60 mg tablet by mouth Daily for 104 weeks
- Placebo IV: Placebo matching with Abatacept injection by intravenous on Days 1,15, 29, and 57, followed by every 4 weeks, Mycophenolate mofetil 1.5 g tablet by mouth and Prednisone up to 60 mg tablet by mouth Daily for 104 Weeks
Period: Year 1 Period
Arm/Group | Abatacept IV | Placebo IV
Started | 203 | 203
Treated | 202 | 203
Completed | 155 (Completed = continued study through Year 1) | 161 (Completed = continued study through Year 1)
Not Completed | 48 | 42
Not completed — Lack of Efficacy | 11 | 9
Not completed — Adverse Event | 20 | 17
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Poor / non-compliance | 0 | 1
Not completed — Pregnancy | 2 | 0
Not completed — Participant no longer meets criteria | 6 | 2
Not completed — Not treated- received ACE inhibition | 1 | 0
Not completed — Change in Concomitant Medication | 0 | 1
Not completed — Need of use of Prohibited Medications | 1 | 0
Not completed — Antiproteinuric changed/dose increased | 0 | 1
Not completed — Hypersensitivity to the medication | 0 | 1
Period: Year 2 Period
Arm/Group | Abatacept IV | Placebo IV
Started | 155 (Started = Completed Year 1) | 161 (Started = Completed Year 1)
Completed | 129 (Completed = Continued study through Year 2) | 123 (Completed = Continued study through Year 2)
Not Completed | 26 | 38
Not completed — Lack of Efficacy | 4 | 12
Not completed — Adverse Event | 7 | 6
Not completed — Participant request to stop treatment | 4 | 4
Not completed — Administrative reason by Sponsor | 4 | 3
Not completed — Participant withdrew consent | 1 | 5
Not completed — Participant no longer meets criteria | 1 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Participant went to US stopped treatment | 0 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Completed Year 1, did not enter Year 2 | 2 | 1
Not completed — Given cyclophosphamide, corticosteroids | 0 | 1
Period: Long-Term Extension (LTE) Period
Arm/Group | Abatacept IV | Placebo IV
Started | 129 (Started = Completed Year 2) | 123 (Started = Completed Year 2)
Completed | 62 (Completed = Continued study through LTE) | 53 (Completed = Continued study through LTE)
Not Completed | 67 | 70
Not completed — Administrative reason by Sponsor | 27 | 21
Not completed — Disease progression | 1 | 4
Not completed — Not effective | 0 | 1
Not completed — Participant request to stop treatment | 1 | 1
Not completed — Participant withdrew consent | 1 | 1
Not completed — Adverse Event unrelated to study drug | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Study drug toxicity | 1 | 0
Not completed — Participant no longer meets criteria | 1 | 0
Not completed — Completed Year 2, did not enter LTE | 33 | 38
Not completed — Absence of renal response | 0 | 1
Not completed — Investigator decision, study termination | 0 | 1
Not completed — Study was terminated | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized and Treated Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept IV | Placebo IV | Total
Number analyzed (Participants) | 202 | 203 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (10.75) [17 to 65] | 33.2 (10.48) [18 to 72] | 33.1 (10.60) [17 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 178 | 360
  Male | 20 | 25 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 71 | 74 | 145
  African American | 15 | 15 | 30
  Caucasian | 85 | 71 | 156
  Other | 31 | 43 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Complete Renal Response (CR) of Lupus Glomerulonephritis at Day 365 of the Double-blind Period
Description: Number of participants achieving CR was divided by the total number of participants in that arm and expressed as a percentage. CR defined as: eGFR is normal or no <85% of the baseline; eGFR based on mean creatinine value from day 358 and 365. Proteinuria: UPCR<0.5 mg/mg. Urine sediment: No cellular casts. Corticosteroid dose: Daily dose must be no >10 mg prednisone or equiv. for at least 28 days prior to assessment. Participants with >10mg/day prednisone or equivalent for non-renal disease within 28 days prior to day 365 will be imputed as having achieved CR if the following are true: Met all criteria for CR at day 337 and all criteria for CR except corticosteroid dose at day 365; Investigator confirms increase in steroid dose is not related to renal disease. Adjusted odds ratio is estimated from logistic regression model which includes treatment group, baseline ACEi/ARBs use (Yes/No), race (Asian/ Black/Caucasian/Other) and baseline UPCR as a continuous variable.
Time Frame: Day 365
Population: All randomized and treated participants
Measure: Number; unit: Percentage
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Percentage | 35.1 [0.8967 to 1.5726] | 33.5
Statistical Analysis 1: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority or Other; p = 0.7264, Stratified logistic regression; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.7077 to 1.6421] — Abatacept IV:Placebo IV 95%CI for Odds Ratio

2. Secondary Outcome: Percentage of Nephrotic Participants in Complete Renal Response of Lupus Glomerulonephritis at Day 365 of the Double-blind Period
Description: Number of participants achieving CR was divided by total participants in that arm, expressed as a percentage. CR is defined the following criteria: eGFR is normal or no <85% of the baseline value; eGFR is based on mean creatinine value from day 358 and 365. Proteinuria: UPCR<0.5 mg/mg. Urine sediment: No cellular casts. Corticosteroid dose: Daily dose must be no >10 mg prednisone or equivalent for at least 28 days prior. Subjects with >10mg/day prednisone or equivalent for non-renal disease within 28 days prior to day 365 will be imputed as CR if the following are true: Met all criteria for CR at day 337 and all criteria for CR except corticosteroid dose at day 365; Investigator confirms increase in steroid dose is not related to renal disease. Adjusted odds ratio is estimated from logistic regression model which includes treatment group, baseline ACEi/ARBs use, race and baseline UPCR as a continuous variable.
Time Frame: Day 365
Population: All randomized and treated nephrotic participants. Nephrotic is defined as screening UPCR >= 3.0mg/mg (>=339mg/mmol)
Measure: Number; unit: Percentage
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 100 | 88
Percentage | 27 [0.8967 to 1.5726] | 29.5
Statistical Analysis 1: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority or Other; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.4148 to 1.5956] — Abatacept IV:Placebo IV

3. Secondary Outcome: Adjusted Mean Change From Baseline in Urine Protein/Creatinine Ratio (UPCR) at Day 365 of the Double-blind Period in Nephrotic Participants
Description: Adjusted Mean Change from Baseline in UPCR at Day 365 of the double-blind period in nephrotic participants
Time Frame: Baseline and Day 365
Population: All randomized and treated nephrotic participants with both post-baseline and baseline measurements
Measure: Mean (Standard Error); unit: UPCR (mg/mg)
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 76 | 68
UPCR (mg/mg) | -5.01 (0.33) | -4.84 (0.35)
Statistical Analysis 1: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis; Adjusted mean difference = -0.17, 95% CI 2-sided [-0.76 to 0.42] — Adjusted mean difference from placebo

4. Secondary Outcome: Adjusted Mean Change From Baseline in UPCR at Day 365 of the Double-blind Period in Overall Population
Description: Adjusted Mean Change from Baseline in Urine protein/creatinine ratio (UPCR) at Day 365 of the double-blind period in the overall population
Time Frame: Day 1 and Day 365
Population: All randomized and treated participants with both post-baseline and baseline measurements
Measure: Mean (Standard Error); unit: UPCR (mg/mg)
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 157 | 163
UPCR (mg/mg) | -2.99 (0.17) | -2.90 (0.16)
Statistical Analysis 1: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority or Other; p = 0.561, Mixed Models Analysis; Adjusted mean difference = -0.09, 95% CI 2-sided [-0.41 to 0.22] — Adjusted mean difference from placebo

5. Secondary Outcome: Adjusted Mean Change From Baseline in Disease Activity as Measured by BILAG 2004 Over Time During Year 1 of the Double-blind Period
Description: Adjusted mean change from baseline in British Isles Lupus Assessment Group (BILAG) score over time during Year 1 of the double-blind period based on a repeated measure mixed model and presented at each visit in the first 12-month of the double-blind period. BILAG index measures disease activity in different organs/systems separately. BILAG score is calculated for each of 9 systems depending on the clinical features present and whether they are new (4 points), worse (3 points), the same (2 points), improving (1 point) or not present (0 points) in the last 4 weeks compared with previously. BILAG "A" represents the presence of serious features of lupus. BILAG "B" represents more moderate features of the disease. BILAG "C" includes only mild symptomatic features. BILAG "D" represents prior activity with no current symptoms due to active lupus. BILAG "E" represents an organ that has never been involved. Overall BILAG score ranges from 0-108, with higher scores reflecting a worse outcome.
Time Frame: Day 1 to Day 365
Population: All randomized and treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 157 | 161
Scores on a Scale | -8.22 [-9.29 to -7.16] | -7.60 [-8.66 to -6.54]

6. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) During Year 1 of the Double-blind Period
Description: All AEs were coded and grouped into preferred terms (PT) by system organ class (SOC), using the Medical Dictionary for Regulatory Activities (MedDRA, version 21.0). Investigators determined the intensity of each AE as mild, moderate, severe, or very severe and assessed the relationship to study drug.
Time Frame: From Day 1 up to 56 days post last dose in Year 1 of the double-blind period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Participants
  Participants with Adverse Events | 188 | 194
  Participants with Serious Adverse Events | 49 | 39
  Participants with infection Adverse Events | 150 | 147
  Participants with malignancies | 2 | 1
  Participants with autoimmune events | 10 | 9
  Participants with peri-infusional Adverse Events | 7 | 9
  Participants with acute infusional Adverse Events | 2 | 4

7. Secondary Outcome: Percentage of Participants With Ranked Outcome of Complete Renal Response, Partial Renal Response (PR), and No Renal Response (NR) During the Double-blind Period
Description: Complete Renal Response or Complete Response (CR): defined as meeting ALL of the following criteria: eGFR normal OR no less than 85% of the baseline value; UPCR < 0.5; Urine sediment: No cellular casts; Daily corticosteroid dose must be no greater than 10 mg prednisone or equivalent for at least 28 days prior to assessment. Partial Renal Response or Partial Response (PR): defined as meeting ALL of the following criteria: Participant does not meet criteria for CR; eGFR no less than 85% of the lesser of the values at screening or randomization (Day 1); UPCR < 0.5 OR 50% reduced from baseline and < 1 if baseline value was < 3, OR 50% reduced from baseline and < 3 if baseline value was greater than or equal to 3; Urine sediment: no cellular casts; daily corticosteroid dose no greater than 10 mg/day prednisone or prednisone equivalent for at least 28 days prior to assessment. No Renal Response or No Response (NR): defined as not meeting criteria for CR or PR or withdrawn
Time Frame: Day 365, Day 729
Population: All randomized and treated participants.
  Year 1 data based on all elements of clinical response definition: UPCR, eGFR and cellular casts.
  Study terminated and Year 2 data based on only two clinical response definition elements: UPCR and eGFR. Data presented for the "as observed" population (those that completed Day 729).
Measure: Number; unit: Percentage
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Percentage
  CR - Day 365 | 35.1 | 33.5
  PR - Day 365 | 20.8 | 21.7
  NR - Day 365 | 44.1 | 44.8
  CR - Day 729: number analyzed (Participants) | 112 | 110
  CR - Day 729 | 60.7 | 53.6
  PR - Day 729: number analyzed (Participants) | 112 | 110
  PR - Day 729 | 25.9 | 22.7
  NR - Day 729: number analyzed (Participants) | 112 | 110
  NR - Day 729 | 13.4 | 23.6
Statistical Analysis 1: Comparison: Abatacept IV vs Placebo IV; CR - Day 365; Test type: Superiority; Estimate of Difference = 1.6510, 95% CI 2-sided [-7.595828 to 10.897784]
Statistical Analysis 2: Comparison: Abatacept IV; PR - Day 365; Test type: Superiority; Estimate of Difference = -0.8828, 95% CI 2-sided [-8.848056 to 7.082461]
Statistical Analysis 3: Comparison: Abatacept IV vs Placebo IV; NR - Day 365; Test type: Superiority; Estimate of Difference = -0.7682, 95% CI 2-sided [-10.446714 to 8.910353]

8. Secondary Outcome: Median Time to Complete Renal Response During the Double-blind Period in All Participants
Description: The estimate of median time to Complete Renal Response is based on Kaplan-Meier analysis. Complete renal response (CR): defined as meeting ALL of the following criteria: eGFR normal OR no less than 85% of the baseline value; Urine protein/creatinine ratio (UPCR) < 0.5; Urine sediment: No cellular casts; Daily corticosteroid dose must be no greater than 10 mg prednisone or equivalent for at least 28 days prior to assessment.
Time Frame: Day 365, Day 729
Population: All randomized and treated participants, as observed, calculated per modified criteria (UPCR and eGFR only)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Days
  Day 365: number analyzed (Participants) | 100 | 98
  Day 365 | 280.0 [198.0 to 365.0] | 309.0 [280.0 to 365.0]
  Day 729: number analyzed (Participants) | 134 | 131
  Day 729 | 170.0 [141.0 to 225.0] | 282.0 [225.0 to 357.0]

9. Secondary Outcome: Median Time to Complete Renal Response During the Double-blind Period in Nephrotic Participants
Description: The estimate of median time to Complete Renal Response in nephrotic participants is based on Kaplan-Meier analysis. Complete renal response (CR): defined as meeting ALL of the following criteria: eGFR normal OR no less than 85% of the baseline value; Urine protein/creatinine ratio (UPCR) < 0.5; Urine sediment: No cellular casts; Daily corticosteroid dose must be no greater than 10 mg prednisone or equivalent for at least 28 days prior to assessment.
Time Frame: Day 365, Day 729
Population: All randomized and treated nephrotic participants, as observed, calculated per modified criteria (UPCR and eGFR only); Nephrotic is defined as screening UPCR >= 3.0 mg/mg (>=339mg/mmol)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 100 | 88
Days
  Day 365: number analyzed (Participants) | 37 | 32
  Day 365 | 366.0 [337.0 to NA] — Study terminated, upper limit not met | 368.0 [311.0 to 368.0]
  Day 729: number analyzed (Participants) | 62 | 51
  Day 729 | 365.0 [197.0 to 644.0] | 368.0 [308.0 to 505.0]

10. Secondary Outcome: Median Time to Partial Renal Response During the Double-blind Period in All Participants
Description: The estimate of median time to Partial Response (PR) is based on Kaplan-Meier analysis. Partial renal response (PR): defined as meeting ALL of the following criteria: Participant does not meet criteria for CR; eGFR no less than 85% of the lesser of the values at screening or randomization (Day 1); UPCR < 0.5 OR 50% reduced from baseline and < 1 if baseline value was < 3, OR 50% reduced from baseline and < 3 if baseline value was 3; Urine sediment: no cellular casts; daily corticosteroid dose no greater than 10 mg/day prednisone or prednisone equivalent for at least 28 days prior to assessment
Time Frame: Day 365, Day 729
Population: All randomized and treated participants, as observed, calculated per modified criteria (UPCR and eGFR only)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Days
  Day 365: number analyzed (Participants) | 105 | 105
  Day 365 | 226.0 [198.0 to 313.0] | 253.0 [198.0 to 358.0]
  Day 729: number analyzed (Participants) | 134 | 131
  Day 729 | 59.0 [56.0 to 85.0] | 58.0 [57.0 to 85.0]

11. Secondary Outcome: Median Time to Partial Renal Response During the Double-blind Period in Nephrotic Participants
Description: The estimate of median time to Partial Response (PR) in nephrotic participants is based on Kaplan-Meier analysis. Partial renal response (PR): defined as meeting ALL of the following criteria: Participant does not meet criteria for CR; eGFR no less than 85% of the lesser of the values at screening or randomization (Day 1); UPCR < 0.5 OR 50% reduced from baseline and < 1 if baseline value was < 3, OR 50% reduced from baseline and < 3 if baseline value was 3; Urine sediment: no cellular casts; daily corticosteroid dose no greater than 10 mg/day prednisone or prednisone equivalent for at least 28 days prior to assessment
Time Frame: Day 365, Day 729
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 100 | 88
Days
  Day 365: number analyzed (Participants) | 55 | 51
  Day 365 | 225.0 [196.0 to 311.0] | 196.0 [170.0 to 225.0]
  Day 729: number analyzed (Participants) | 62 | 51
  Day 729 | 58.5 [29.0 to 86.0] | 56.0 [29.0 to 58.0]

12. Secondary Outcome: Adjusted Mean Change From Baseline in UPCR Over Time
Description: A repeated measure mixed model that included the baseline UPCR value, randomization stratification factors, time, and time by treatment interaction as fixed effects and subject as a random effect was used.
Time Frame: Day 365; Day 729, includes data up to July 1st 2017 when double-blind therapy ended
Population: All randomized and treated participants with both post-baseline and baseline measurements
Measure: Mean (Standard Error); unit: UPCR (mg/mg)
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 157 | 163
UPCR (mg/mg)
  Day 365 | -2.95 (0.17) | -2.68 (0.17)
  Day 729: number analyzed (Participants) | 112 | 110
  Day 729 | -3.13 (0.18) | -2.72 (0.18)

13. Secondary Outcome: Median Percent Change From Baseline in UPCR Over Time
Description: A repeated measure mixed model that included the baseline UPCR value, randomization stratification factors, time, and time by treatment interaction as fixed effects and subject as a random effect was used.
  % Change from Baseline = (post baseline - baseline value) / baseline value x 100
Time Frame: Day 365, Day 729
Population: All randomized and treated participants with both post-baseline and baseline measurements
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Percent
  Day 365: number analyzed (Participants) | 157 | 163
  Day 365 | -83.77 [-92.42 to -64.18] | -84.12 [-94.03 to -59.98]
  Day 729: number analyzed (Participants) | 112 | 110
  Day 729 | -89.83 [-95.41 to -77.95] | -87.28 [-93.78 to -66.43]

14. Secondary Outcome: Adjusted Mean Change From Baseline in eGFR Over Time
Description: Estimated glomerular filtration rate(eGFR), will be calculated by the CKD-EPI formula shown below.50 eGFR is expressed as mL/min per 1.73m2. For the purpose of this study lower limit of normal eGFR is defined as 90mL/min per 1.73m2 eGFR = 141 X min (Scr/k, 1)α X max (Scr/k, 1)-1.209 X 0.993Age X (1.018 [if female]) X (1.159 [if black]) Where Scr is serum creatinine (mg/dL), k is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1, age in years.
Time Frame: Day 365, Day 729
Population: All randomized and treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: mL/min per 1.73m2
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
mL/min per 1.73m2
  Day 365: number analyzed (Participants) | 158 | 162
  Day 365 | 6.85 [3.47 to 10.23] | 5.85 [2.51 to 9.20]
  Day 729: number analyzed (Participants) | 112 | 109
  Day 729 | 7.20 [3.40 to 11.00] | 7.91 [4.14 to 11.68]

15. Secondary Outcome: Median Time to First Sustained Change to No Response During the Double-blind Period
Description: Sustained response defined as response present at 2 consecutive visits approximately 4 weeks apart. No renal response (NR): defined as not meeting criteria for CR or PR or withdrawn
  The estimate of median time is based on Kaplan-Meier analysis
Time Frame: Day 365, Day 729
Population: All randomized and treated participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Days
  Day 365: number analyzed (Participants) | 23 | 19
  Day 365 | NA [392.0 to NA] — Due to < 50% event occurrence, the median is not evaluable | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable
  Day 729 | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable | NA [672.0 to NA] — Due to < 50% event occurrence, the median is not evaluable

16. Secondary Outcome: Number of Participants With Sustained Change From Higher Level of Response to no Response During the Double-blind Period
Description: Sustained change to no response is defined as going from CR (or PR) to NR and remaining in NR for at least 2 consecutive visits; visits should be approximately 4 weeks apart. This analysis will be based on time from response CR (or PR) to the first visit in which the no response (NR) was achieved and sustained to the next visit.
Time Frame: Day 365, Day 729
Population: All randomized and treated participants, as observed, calculated per modified criteria (UPCR and eGFR only)
Measure: Number; unit: Participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Participants
  Day 365: number analyzed (Participants) | 110 | 98
  Day 365 | 5 | 3
  Day 729: number analyzed (Participants) | 134 | 131
  Day 729 | 52 | 56
Statistical Analysis 1: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority — Day 365; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.3251 to 6.2849]
Statistical Analysis 2: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority — Day 729; Estimate of Difference vs Drug = 3.4, 95% CI 2-sided [-8.4 to 15.1]

17. Secondary Outcome: Adjusted Mean Change From Baseline in Disease Activity as Measured by BILAG 2004 Over Time During the Double-blind Period
Description: BILAG index measures and reports disease activity in different organs/systems separately. The BILAG score is calculated for each of nine systems depending on the clinical features present and whether they are new (4 points), worse (3 points), the same (2 points), improving (1 point) or not present (0 points) in the last 4 weeks compared with previously. A BILAG "A" represents the presence of one or more serious features of lupus. A BILAG "B" represents more moderate features of the disease. A BILAG "C" includes only mild symptomatic features. A BILAG "D" represents only prior activity with no current symptoms due to active lupus. A BILAG "E" represents an organ that has never been involved. Overall BILAG score ranges from 0-108, with higher scores reflecting a worse outcome.
Time Frame: Day 1 to Day 729; Day 365 to Day 729
Population: All randomized and treated participants with both post-baseline and baseline measurements
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Scores on a Scale
  Day 1 to Day 729: number analyzed (Participants) | 109 | 108
  Day 1 to Day 729 | -9.31 (0.56) | -8.53 (0.56)
  Day 365 to Day 729: number analyzed (Participants) | 129 | 127
  Day 365 to Day 729 | -0.95 (0.538) | -0.40 (0.530)

18. Secondary Outcome: Cmin (ug/mL): Trough Level Serum Concentration of Abatacept Prior to the Administration of the IV Infusion
Description: Trough level serum concentration of abatacept prior to the administration of the IV infusion on Days 1 to 365
Time Frame: Days 1 to 365
Population: All participants who received at least 1 Abatacept Infusion and have at least 1 Cmin value during Year 1 of the double-blind period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 189 | 0
ug/mL
  Day 15 | 69.97 (91.4) |
  Day 29: number analyzed (Participants) | 177 | 0
  Day 29 | 90.46 (56.8) |
  Day 57: number analyzed (Participants) | 177 | 0
  Day 57 | 36.43 (84.4) |
  Day 85: number analyzed (Participants) | 172 | 0
  Day 85 | 34.46 (55.4) |
  Day 113: number analyzed (Participants) | 164 | 0
  Day 113 | 16.42 (69.2) |
  Day 169: number analyzed (Participants) | 157 | 0
  Day 169 | 13.98 (64.5) |
  Day 281: number analyzed (Participants) | 152 | 0
  Day 281 | 14.44 (54.7) |
  Day 337: number analyzed (Participants) | 139 | 0
  Day 337 | 14.99 (73.6) |
  Day 365: number analyzed (Participants) | 133 | 0
  Day 365 | 13.62 (51.7) |

19. Secondary Outcome: Cmax: Maximum Observed Serum Concentration Following Participants Receiving Active Abatacept IV
Description: Cmax: Maximum observed serum concentration following participants receiving active abatacept IV
Time Frame: at 1 hour post Day 1 dose and 30 minutes post Day 337 dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 185 | 0
ug/mL
  Day 1 | 527.43 (59.6) |
  Day 337: number analyzed (Participants) | 135 | 0
  Day 337 | 203.51 (30.6) |

20. Secondary Outcome: AUC (TAU): Area Under the Serum Concentration Time Curve Over a Dosing Interval
Description: AUC (TAU): Area under the serum concentration time curve over a dosing interval between Days 337 to 365.
Time Frame: Days 337 to 365
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 106 | 0
ug*h/mL | 36480.24 (29.2) |

21. Secondary Outcome: Summary Statistics for Systolic Blood Pressure
Description: Summary statistics for systolic blood pressure
Time Frame: Day 1 to Day 729
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
mmHg
  Day 1, end of observation: number analyzed (Participants) | 199 | 200
  Day 1, end of observation | 122.0 (15.48) | 122.6 (15.31)
  Day 365, end of observation: number analyzed (Participants) | 4 | 2
  Day 365, end of observation | 112.3 (18.45) | 115.0 (7.07)
  Day 729, end of observation: number analyzed (Participants) | 81 | 73
  Day 729, end of observation | 108.6 (13.29) | 114.2 (14.51)

22. Secondary Outcome: Summary Statistics for Diastolic Blood Pressure
Description: Summary statistics for diastolic blood pressure
Time Frame: Day 1 to Day 729
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
mmHg
  Day 1, end of observation: number analyzed (Participants) | 199 | 200
  Day 1, end of observation | 76.5 (11.49) | 77.0 (11.19)
  Day 365, end of observation: number analyzed (Participants) | 4 | 2
  Day 365, end of observation | 73.5 (10.75) | 77.5 (10.61)
  Day 729, end of observation: number analyzed (Participants) | 81 | 73
  Day 729, end of observation | 67.5 (9.60) | 72.7 (9.45)

23. Secondary Outcome: Summary Statistics for Heart Rate
Description: Summary statistics for Heart Rate
Time Frame: Day 1 to Day 729
Population: All treated participants
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
beats per minute
  Day 1, end of observation: number analyzed (Participants) | 199 | 200
  Day 1, end of observation | 80.6 (10.91) | 81.4 (10.64)
  Day 365, end of observation: number analyzed (Participants) | 4 | 2
  Day 365, end of observation | 78.5 (9.57) | 70.0 (14.14)
  Day 729, end of observation: number analyzed (Participants) | 81 | 72
  Day 729, end of observation | 76.2 (11.69) | 76.7 (10.36)

24. Secondary Outcome: Mean Change From Baseline in Laboratory Analytes During the Double-blind Period (U/L)
Description: Laboratory assessments were analyzed centrally, with the exception of pregnancy testing. Blood draws and urine collections were performed at visits specified in the protocol.
  Change from Baseline = Post-baseline - Baseline value.
Time Frame: Day 729
Population: All treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
U/L
  ALANINE AMINOTRANSFERASE (ALT) (U/L): number analyzed (Participants) | 133 | 116
  ALANINE AMINOTRANSFERASE (ALT) (U/L) | -2.2 [-4.834 to 0.382] | -3.4 [-6.462 to -0.435]
  ALKALINE PHOSPHATASE (ALP) (U/L): number analyzed (Participants) | 133 | 116
  ALKALINE PHOSPHATASE (ALP) (U/L) | 8.2 [4.514 to 11.967] | 11.7 [7.125 to 16.202]
  ASPARTATE AMINOTRANSFERASE (AST) (U/L): number analyzed (Participants) | 133 | 116
  ASPARTATE AMINOTRANSFERASE (AST) (U/L) | 0.3 [-1.747 to 2.288] | 0.3 [-1.326 to 1.947]
  G-GLUTAMYL TRANSFERASE (GGT) (U/L): number analyzed (Participants) | 133 | 116
  G-GLUTAMYL TRANSFERASE (GGT) (U/L) | -5.3 [-11.020 to 0.509] | -4.1 [-11.419 to 3.143]

25. Secondary Outcome: Mean Change From Baseline in Laboratory Analytes During the Double-blind Period (g/L)
Description: as for outcome 24
Time Frame: Day 729
Population: All treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: g/L
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
g/L
  ALBUMIN (g/L): number analyzed (Participants) | 133 | 116
  ALBUMIN (g/L) | 9.2 [8.040 to 10.336] | 8.1 [6.917 to 9.308]
  HEMOGLOBIN (g/L): number analyzed (Participants) | 129 | 113
  HEMOGLOBIN (g/L) | 8.8 [5.977 to 11.574] | 9.0 [5.480 to 12.449]
  PROTEIN, TOTAL (g/L) | 9.9 [8.135 to 11.579] | 10.1 [8.438 to 11.786]

26. Secondary Outcome: Mean Change From Baseline in Laboratory Analytes During the Double-blind Period (Percentage of Blood)
Description: as for outcome 24
Time Frame: Day 729
Population: All treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
Percentage | 0.0328 [0.023873 to 0.041658] | 0.0325 [0.021813 to 0.043160]

27. Secondary Outcome: Mean Change From Baseline in Laboratory Analytes During the Double-blind Period (Umol/L)
Description: as for outcome 24
Time Frame: Day 729
Population: All treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
umol/L
  BILIRUBIN, TOTAL (umol/L): number analyzed (Participants) | 133 | 116
  BILIRUBIN, TOTAL (umol/L) | 1.77 [1.0751 to 2.4633] | 1.00 [0.5112 to 1.4922]
  CREATININE (umol/L): number analyzed (Participants) | 133 | 116
  CREATININE (umol/L) | -5.6 [-9.306 to -1.912] | -6.2 [-10.764 to -1.598]

28. Secondary Outcome: Mean Change From Baseline in Laboratory Analytes During the Double-blind Period (mmol/L)
Description: as for outcome 24
Time Frame: Day 729
Population: All treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
mmol/L
  BLOOD UREA NITROGEN (mmol/L): number analyzed (Participants) | 133 | 116
  BLOOD UREA NITROGEN (mmol/L) | -2.31 [-2.9879 to -1.6241] | -2.25 [-2.8370 to -1.6682]
  CALCIUM, TOTAL (mmol/L): number analyzed (Participants) | 133 | 116
  CALCIUM, TOTAL (mmol/L) | 0.097 [0.06893 to 0.12566] | 0.108 [0.07754 to 0.13850]
  CHLORIDE, SERUM (mmol/L): number analyzed (Participants) | 133 | 116
  CHLORIDE, SERUM (mmol/L) | -1.1 [-1.675 to -0.461] | -0.5 [-1.244 to 0.192]
  GLUCOSE, SERUM (mmol/L): number analyzed (Participants) | 116 | 101
  GLUCOSE, SERUM (mmol/L) | -0.23 [-0.4924 to 0.0424] | -0.58 [-0.9623 to -0.1902]
  PHOSPHORUS, INORGANIC (mmol/L): number analyzed (Participants) | 133 | 116
  PHOSPHORUS, INORGANIC (mmol/L) | -0.077 [-0.12699 to -0.02654] | -0.037 [-0.08152 to 0.00807]
  POTASSIUM, SERUM (mmol/L) | -0.02 [-0.0947 to 0.0646] | -0.10 [-0.2115 to 0.0029]
  SODIUM, SERUM (mmol/L) | -0.2 [-0.762 to 0.280] | -0.5 [-1.060 to 0.078]

29. Secondary Outcome: Mean Change From Baseline in Laboratory Analytes During the Double-blind Period (x10^9 Cells/L)
Description: as for outcome 24
Time Frame: Day 729
Population: All treated participants with both post-baseline and baseline measurements
Measure: Mean (95% Confidence Interval); unit: x10^9 cells/L
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
x10^9 cells/L
  EOSINOPHILS (ABSOLUTE) (x10^9 cells/L): number analyzed (Participants) | 126 | 113
  EOSINOPHILS (ABSOLUTE) (x10^9 cells/L) | 0.034 [0.01182 to 0.05611] | 0.010 [-0.01781 to 0.03781]
  LYMPHOCYTES (ABSOLUTE) (x10^9 cells/L): number analyzed (Participants) | 126 | 113
  LYMPHOCYTES (ABSOLUTE) (x10^9 cells/L) | 0.141 [-0.01315 to 0.29584] | -0.149 [-0.29961 to 0.00138]
  MONOCYTES (ABSOLUTE) (x10^9 cells/L): number analyzed (Participants) | 126 | 113
  MONOCYTES (ABSOLUTE) (x10^9 cells/L) | -0.018 [-0.05220 to 0.01649] | -0.050 [-0.09264 to -0.00772]
  NEUTROPHILS (ABSOLUTE) (x10^9 cells/L): number analyzed (Participants) | 126 | 113
  NEUTROPHILS (ABSOLUTE) (x10^9 cells/L) | -2.259 [-2.78568 to -1.73210] | -2.289 [-2.95652 to -1.62118]
  PLATELET COUNT (x10^9 cells/L): number analyzed (Participants) | 129 | 112
  PLATELET COUNT (x10^9 cells/L) | -4.9 [-16.962 to 7.148] | -9.1 [-24.094 to 5.951]

30. Secondary Outcome: Number of Participants With Marked Hematology Laboratory Abnormalities During Year 1 of the Double Blind Period
Description: LLN= Lower limit of normals ULN= Upper limit of normals Pre RX = Baseline value HEMOGLOBIN g/L 4.0 HB >3 G/DL DECREASE FROM PRE RX HEMATOCRIT vol 6.3 HCT <0.75X PRE RX ERYTHROCYTES x10*12 c/L 5.2 RBC <0.75X PRE RX PLATELET COUNT x10*9 c/L 5.0 PLAT <0.67X LLN OR >1.5X ULN, OR IF PRE RX<LLN THEN USE 0.5X PRE RX AND <100,000/MM3 LEUKOCYTES x10*9 c/L 6.2 WBC <0.75X LLN OR >1.25X ULN, OR IF PRE RX<LLN THEN USE <0.8X PRE RX OR >ULN, OR IF PRE RX>ULN THEN USE >1.2X PRE RX OR <LLN EOSINOPHILS (ABSOLUTE) x10*9 c/L 8.3 EOSA IF VALUE > .750 X10*3 c/uL BASOPHILS (ABSOLUTE) x10*9 c/L 8.3 BASOA IF VALUE > 400/MM3 MONOCYTES (ABSOLUTE) x10*9 c/L 8.3 MONOA IF VALUE > 2000/MM3 LYMPHOCYTES (ABSOLUTE) x10*9 c/L 8.3 LYMPA IF VALUE < .750 X10*3 c/uL OR IF VALUE > 7.50 X10*3 c/uL
  N = the number of participants with at least 1 on treatment lab result for each analyte
Time Frame: Day 1 to Day 365; includes data up to 56 days post last dose in year 1 of double-blind period or first dose date in the year 2 of double-blind period, whichever is earlier
Population: All treated participants
  NA (not available) indicates not-calculated as it was not a relevant pre-specified marked abnormality.
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
participants
  HEMOGLOBIN, low | 6 | 10
  HEMOGLOBIN, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  HEMATOCRIT, low: number analyzed (Participants) | 201 | 203
  HEMATOCRIT, low | 12 | 12
  HEMATOCRIT, high: number analyzed (Participants) | 201 | 203
  HEMATOCRIT, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ERYTHROCYTES, low: number analyzed (Participants) | 201 | 203
  ERYTHROCYTES, low | 7 | 10
  ERYTHROCYTES, high: number analyzed (Participants) | 201 | 203
  ERYTHROCYTES, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  PLATELET COUNT, low: number analyzed (Participants) | 201 | 203
  PLATELET COUNT, low | 4 | 3
  PLATELET COUNT, high: number analyzed (Participants) | 201 | 203
  PLATELET COUNT, high | 0 | 0
  LEUKOCYTES, low | 35 | 21
  LEUKOCYTES, high | 29 | 25
  EOSINOPHILS (ABSOLUTE), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  EOSINOPHILS (ABSOLUTE), high | 2 | 6
  BASOPHILS (ABSOLUTE), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BASOPHILS (ABSOLUTE), high | 1 | 1
  MONOCYTES (ABSOLUTE), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  MONOCYTES (ABSOLUTE), high | 0 | 1
  LYMPHOCYTES (ABSOLUTE), low | 81 | 104
  LYMPHOCYTES (ABSOLUTE), high | 1 | 2

31. Secondary Outcome: Number of Participants With Marked Liver and Kidney Function Laboratory Abnormalities During Year 1 of the Double Blind Period
Description: LLN= Lower limit of normals ULN= Upper limit of normals Pre RX = Baseline value ALKALINE PHOSPHATASE (ALP) U/L 5.0 ALP >2X ULN, OR IF PRE RX>ULN THEN USE >3X PRE RX ASPARTATE AMINOTRANSFERASE (AST) U/L 5.0 AST >3X ULN, OR IF PRE RX>ULN THEN USE >4X PRE RX ALANINE AMINOTRANSFERASE (ALT) U/L 5.0 ALT >3X ULN, OR IF PRE RX>ULN THEN USE >4X PRE RX G-GLUTAMYL TRANSFERASE (GGT) U/L 5.0 GGT >2X ULN, OR IF PRE RX>ULN THEN USE >3X PRE RX BILIRUBIN, TOTAL umol/L 5.1 TBILI >2X ULN, OR IF PRE RX>ULN THEN USE >4X PRE RX BILIRUBIN, DIRECT umol/L 5.1 DBILI >1.5X ULN, OR IF PRE RX>ULN THEN USE >2X PRE RX BLOOD UREA NITROGEN mmol/L 5.1 BUN >2X PRE RX CREATININE umol/L 5.0 CREAT >1.5X PRE RX
  N = the number of participants with at least 1 on treatment lab result for each analyte
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
participants
  ALKALINE PHOSPHATASE (ALP), low: number analyzed (Participants) | 201 | 203
  ALKALINE PHOSPHATASE (ALP), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ALKALINE PHOSPHATASE (ALP), high: number analyzed (Participants) | 201 | 203
  ALKALINE PHOSPHATASE (ALP), high | 1 | 1
  ASPARTATE AMINOTRANSFERASE (AST), low: number analyzed (Participants) | 201 | 203
  ASPARTATE AMINOTRANSFERASE (AST), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ASPARTATE AMINOTRANSFERASE (AST), high: number analyzed (Participants) | 201 | 203
  ASPARTATE AMINOTRANSFERASE (AST), high | 5 | 0
  ALANINE AMINOTRANSFERASE (ALT), low: number analyzed (Participants) | 201 | 203
  ALANINE AMINOTRANSFERASE (ALT), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ALANINE AMINOTRANSFERASE (ALT), high: number analyzed (Participants) | 201 | 203
  ALANINE AMINOTRANSFERASE (ALT), high | 8 | 2
  G-GLUTAMYL TRANSFERASE (GGT), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  G-GLUTAMYL TRANSFERASE (GGT), high | 17 | 15
  BILIRUBIN, TOTAL, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BILIRUBIN, TOTAL, high | 0 | 0
  BILIRUBIN, DIRECT, low: number analyzed (Participants) | 200 | 203
  BILIRUBIN, DIRECT, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BILIRUBIN, DIRECT, high: number analyzed (Participants) | 200 | 203
  BILIRUBIN, DIRECT, high | 0 | 0
  BLOOD UREA NITROGEN, low: number analyzed (Participants) | 201 | 203
  BLOOD UREA NITROGEN, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BLOOD UREA NITROGEN, high: number analyzed (Participants) | 201 | 203
  BLOOD UREA NITROGEN, high | 20 | 12
  CREATININE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  CREATININE, high | 24 | 20

32. Secondary Outcome: Number of Participants With Marked Electrolyte Laboratory Abnormalities During Year 1 of the Double Blind Period
Description: LLN= Lower limit of normals ULN= Upper limit of normals Pre RX = Baseline value SODIUM, SERUM mmol/L 4.0 NA <0.95X LLN OR >1.05X ULN, OR IF PRE RX<LLN THEN USE <0.95X PRE RX OR >ULN, OR IF PRE RX>ULN THEN USE >1.05X PRE RX OR <LLN POTASSIUM, SERUM mmol/L 4.1 K <0.9X LLN OR >1.1X ULN, OR IF PRE RX<LLN THEN USE <0.9X PRE RX OR >ULN, OR IF PRE RX>ULN THEN USE >1.1X PRE RX OR <LLN CHLORIDE, SERUM mmol/L 5.0 CL <0.9X LLN OR >1.1X ULN, OR IF PRE RX<LLN THEN USE <0.9X PRE RX OR >ULN, OR IF PRE RX>ULN THEN USE >1.1X PRE RX OR <LLN
  N = the number of participants with at least 1 on treatment lab result for each analyte
Time Frame: as for outcome 30
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
participants
  SODIUM, SERUM, low | 1 | 1
  SODIUM, SERUM, high | 2 | 2
  POTASSIUM, SERUM, low | 3 | 5
  POTASSIUM, SERUM, high | 7 | 7
  CHLORIDE, SERUM, low | 0 | 1
  CHLORIDE, SERUM, high | 0 | 0
  CALCIUM, TOTAL, low | 1 | 1
  CALCIUM, TOTAL, high | 2 | 0
  PHOSPHORUS, INORGANIC, low | 9 | 7
  PHOSPHORUS, INORGANIC, high | 13 | 13

33. Secondary Outcome: Number of Participants With Marked Urinalysis Laboratory Abnormalities During Year 1 of the Double Blind Period
Description: LLN= Lower limit of normals ULN= Upper limit of normals Pre RX = Baseline value PROTEIN, URINE Unknown UPRO IF MISSING PRE THEN USE >=2, OR IF VALUE >=4, OR IF PRE RX =0 OR 0.5 THEN USE >=2, OR IF PRE RX =1 THEN USE >=3, OR IF PRE RX =2 OR 3 THEN USE >=4 GLUCOSE, URINE N/A UGLU IF MISSING PRE THEN USE >=2, OR IF VALUE >=4, OR IF PRE RX =0 OR 0.5 THEN USE >=2, OR IF PRE RX =1 THEN USE >=3, OR IF PRE RX =2 OR 3 THEN USE >=4 BLOOD, URINE N/A UBLD IF MISSING PRE THEN USE >=2, OR IF VALUE >=4, OR IF PRE RX =0 OR 0.5 THEN USE >=2, OR IF PRE RX =1 THEN USE >=3, OR IF PRE RX =2 OR 3 THEN USE >=4 RBC, URINE hpf 5.0 URBC IF MISSING PRE THEN USE >=2, OR IF VALUE >=4, OR IF PRE RX =0 OR 0.5 THEN USE >=2, OR IF PRE RX =1 THEN USE >=3, OR IF PRE RX =2 OR 3 THEN USE >=4 WBC, URINE hpf 5.0 UWBC IF MISSING PRE THEN USE >=2, OR IF VALUE >=4, OR IF PRE RX =0 OR 0.5 THEN USE >=2, OR IF PRE RX =1 THEN USE >=3, OR IF PRE RX =2 OR 3 THEN USE >=4
Time Frame: as for outcome 30
Population: All treated participants
  N = the number of participants with at least 1 on treatment lab result for each analyte
  NA (not available) indicates not-calculated as it was not a relevant pre-specified marked abnormality.
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
participants
  PROTEIN, URINE, low: number analyzed (Participants) | 198 | 195
  PROTEIN, URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  PROTEIN, URINE, high: number analyzed (Participants) | 198 | 195
  PROTEIN, URINE, high | 0 | 0
  GLUCOSE, URINE, low: number analyzed (Participants) | 193 | 194
  GLUCOSE, URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  GLUCOSE, URINE, high: number analyzed (Participants) | 193 | 194
  GLUCOSE, URINE, high | 0 | 0
  BLOOD, URINE, low: number analyzed (Participants) | 200 | 200
  BLOOD, URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BLOOD, URINE, high: number analyzed (Participants) | 200 | 200
  BLOOD, URINE, high | 0 | 0
  Red blood cells (RBC), URINE, low: number analyzed (Participants) | 201 | 201
  Red blood cells (RBC), URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  Red blood cells (RBC), URINE, high: number analyzed (Participants) | 201 | 201
  Red blood cells (RBC), URINE, high | 93 | 103
  White blood cells (WBC), URINE, low: number analyzed (Participants) | 201 | 201
  White blood cells (WBC), URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  White blood cells (WBC), URINE, high: number analyzed (Participants) | 201 | 201
  White blood cells (WBC), URINE, high | 91 | 98

34. Secondary Outcome: Number of Participants With Other Marked Chemistry Laboratory Abnormalities During Year 1 of the Double Blind Period
Description: LLN= Lower limit of normals ULN= Upper limit of normals Pre RX = Baseline value CALCIUM, TOTAL mmol/L 5.2 CA <0.8X LLN OR >1.2X ULN, OR IF PRE RX<LLN THEN USE <0.75X PRE RX OR >ULN, OR IF PRE RX>ULN THEN USE >1.25X PRE RX OR <LLN PHOSPHORUS, INORGANIC mmol/L 5.2 PHOS <0.75X LLN OR >1.25X ULN, OR IF PRE RX<LLN THEN USE <0.67X PRE RX OR >ULN GLUCOSE, SERUM mmol/L 4.1 GLUC <65 mg/dL, OR >220 mg/dL PROTEIN, TOTAL g/L 5.0 TPRO <0.9X LLN OR >1.1X ULN, OR IF PRE RX<LLN THEN USE 0.9X PRE RX OR >ULN, OR IF PRE RX>ULN THEN USE 1.1X PRE RX OR <LLN ALBUMIN g/L 3.0 ALB <0.9X LLN, OR IF PRE RX<LLN THEN USE <0.75X PRE RX CHOLESTEROL, TOTAL (TC) mmol/L 5.2 CHOL >2X PRE R
  N = the number of participants with at least 1 on treatment lab result for each analyte
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
participants
  GLUCOSE, SERUM, low | 33 | 29
  GLUCOSE, SERUM, high | 10 | 5
  PROTEIN, TOTAL, low: number analyzed (Participants) | 201 | 203
  PROTEIN, TOTAL, low | 44 | 26
  PROTEIN, TOTAL, high: number analyzed (Participants) | 201 | 203
  PROTEIN, TOTAL, high | 0 | 1
  ALBUMIN, low | 10 | 11
  ALBUMIN, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value

35. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) During Year 2 of the Double-blind Period and Long-term Extension
Description: as for outcome 6
Time Frame: From the first dose in Year 2 of the double-blind period up to 56 days post last dose
Population: All treated participants in Year 2
Measure: Number; unit: Participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
Participants
  Participants with Adverse Events | 127 | 137
  Participants with Serious Adverse Events | 15 | 25
  Participants with infection Adverse Events | 100 | 107
  Participants with malignancies | 0 | 1
  Participants with autoimmune events | 7 | 11

36. Secondary Outcome: Percentage of Participants in Treatment Failure Over Time During the Double-blind Period
Description: Lupus treatment failure is defined as any of the following: Death, unless due to physical trauma or violence; Renal Flare; sustained doubling of creatinine from baseline (greater of Screening or Study Day 1 value); initiation of rescue therapy for treatment of active lupus nephritis after Study Week 20.
  Overall treatment failure is defined as lupus treatment failure plus discontinuation of study drug for any reason except death due to physical trauma or violence, pregnancy or administrative decision by Sponsor.
Time Frame: Day 365, Day 729
Population: All randomized and treated participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Percentage
  Lupus treatment failure (LTF) - Day 365 | 3.5 [0.943 to 5.988] | 4.4 [1.602 to 7.265]
  Overall treatment failure (OTF) - Day 365 | 4.5 [1.610 to 7.301] | 4.9 [1.949 to 7.903]
  LTF - Day 729: number analyzed (Participants) | 134 | 131
  LTF - Day 729 | 4.5 [1.0 to 8.0] | 5.3 [1.5 to 9.2]
  OTF - Day 729: number analyzed (Participants) | 134 | 131
  OTF - Day 729 | 5.2 [1.5 to 9.0] | 8.4 [3.6 to 13.1]
Statistical Analysis 1: Comparison: Abatacept IV vs Placebo IV; Lupus treatment failure - Day 365; Test type: Superiority; Estimate of Difference = -0.9682, 95% CI 2-sided [-4.760178 to 2.823876]
Statistical Analysis 2: Comparison: Abatacept IV; Overall treatment failure - Day 365; Test type: Superiority; Estimate of Difference = -0.4707, 95% CI 2-sided [-4.588691 to 3.647365]
Statistical Analysis 3: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority — Lupus treatment failure - Day 729; Estimate of Difference = 0.8, 95% CI 2-sided [-4.5 to 6.1]
Statistical Analysis 4: Comparison: Abatacept IV vs Placebo IV; Test type: Superiority — Overall treatment failure - Day 729; Estimate of Difference = 2.7, 95% CI 2-sided [-3.3 to 8.8]

37. Secondary Outcome: Median Time to First Treatment Failure and Overall Treatment Failure During the Double-blind Period
Description: First treatment failure (or Lupus treatment failure) is defined as any of the following: Death, unless due to physical trauma or violence; Renal Flare; sustained doubling of creatinine from baseline (greater of Screening or Study Day 1 value); initiation of rescue therapy for treatment of active lupus nephritis after Study Week 20.
  Overall treatment failure is defined as lupus treatment failure plus discontinuation of study drug for any reason except death due to physical trauma or violence, pregnancy or administrative decision by Sponsor.
  The hazard ratio is estimated using the Cox proportional hazards model which includes treatment group, stratification variables (baseline ACEis/ARBs use, RACE) and baseline UPCR.
  The estimate of median time is based on Kaplan-Meier analysis
Time Frame: Day 365, Day 729
Population: All randomized and treated participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Days
  First treatment failure (FTF) - Day 365: number analyzed (Participants) | 56 | 50
  First treatment failure (FTF) - Day 365 | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable
  Overall treatment failure (OTF) - Day 365: number analyzed (Participants) | 74 | 71
  Overall treatment failure (OTF) - Day 365 | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable
  FTF - Day 729 | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable
  OTF - Day 729 | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable | NA [NA to NA] — Due to < 50% event occurrence, the median is not evaluable

38. Secondary Outcome: Percentage of Nephrotic Participants in Complete Renal Response of Lupus Glomerulonephritis at Day 729 of the Double-blind Period
Description: as for outcome 2
Time Frame: Day 729
Population: All randomized and treated nephrotic participants, as observed, calculated per modified criteria (UPCR and eGFR only). Nephrotic is defined as screening UPCR >= 3.0mg/mg (>=339mg/mmol)
Measure: Number; unit: Percentage
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 62 | 51
Percentage | 50.0 | 49.0

39. Secondary Outcome: Percentage of Participants in Overall Population in Complete Renal Response of Lupus Glomerulonephritis at Day 729 of the Double-blind Period
Description: as for outcome 2
Time Frame: Day 729
Population: All randomized and treated participants, as observed, calculated per modified criteria (UPCR and eGFR only)
Measure: Number; unit: Percentage
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 134 | 131
Percentage | 61.9 | 52.7

40. Secondary Outcome: Number of Participants With Marked Hematology Laboratory Abnormalities in the Double Blind Period
Description: as for outcome 30
Time Frame: Day 1 to Day 729
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
participants
  HEMOGLOBIN, low | 8 | 9
  HEMOGLOBIN, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  HEMATOCRIT, low | 6 | 2
  HEMATOCRIT, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ERYTHROCYTES, low | 4 | 2
  ERYTHROCYTES, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  PLATELET COUNT, low | 2 | 4
  PLATELET COUNT, high | 1 | 0
  LEUKOCYTES, low | 19 | 24
  LEUKOCYTES, high | 3 | 5
  EOSINOPHILS (ABSOLUTE), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  EOSINOPHILS (ABSOLUTE), high | 11 | 6
  BASOPHILS (ABSOLUTE), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BASOPHILS (ABSOLUTE), high | 0 | 0
  MONOCYTES (ABSOLUTE), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  MONOCYTES (ABSOLUTE), high | 0 | 0
  LYMPHOCYTES (ABSOLUTE), low | 43 | 62
  LYMPHOCYTES (ABSOLUTE), high | 0 | 0

41. Secondary Outcome: Number of Participants With Marked Liver and Kidney Function Laboratory Abnormalities in the Double Blind Period
Description: as for outcome 31
Time Frame: Day 1 to Day 729
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
participants
  ALKALINE PHOSPHATASE (ALP), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ALKALINE PHOSPHATASE (ALP), high | 4 | 0
  ASPARTATE AMINOTRANSFERASE (AST), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ASPARTATE AMINOTRANSFERASE (AST), high | 2 | 3
  ALANINE AMINOTRANSFERASE (ALT), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  ALANINE AMINOTRANSFERASE (ALT), high | 4 | 3
  G-GLUTAMYL TRANSFERASE (GGT), low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  G-GLUTAMYL TRANSFERASE (GGT), high | 17 | 11
  BILIRUBIN, TOTAL, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BILIRUBIN, TOTAL, high | 0 | 0
  BILIRUBIN, DIRECT, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BILIRUBIN, DIRECT, high | 1 | 0
  BLOOD UREA NITROGEN, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BLOOD UREA NITROGEN, high | 10 | 9
  CREATININE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  CREATININE, high | 17 | 16

42. Secondary Outcome: Number of Participants With Marked Electrolyte Laboratory Abnormalities in the Double Blind Period
Description: as for outcome 32
Time Frame: Day 1 to Day 729
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
participants
  SODIUM, SERUM, low | 0 | 0
  SODIUM, SERUM, high | 0 | 1
  POTASSIUM, SERUM, low | 2 | 2
  POTASSIUM, SERUM, high | 3 | 2
  CHLORIDE, SERUM, low | 0 | 1
  CHLORIDE, SERUM, high | 0 | 0
  CALCIUM, TOTAL, low | 0 | 0
  CALCIUM, TOTAL, high | 1 | 0
  PHOSPHORUS, INORGANIC, low | 3 | 4
  PHOSPHORUS, INORGANIC, high | 6 | 3

43. Secondary Outcome: Number of Participants With Marked Urinalysis Laboratory Abnormalities in the Double Blind Period
Description: as for outcome 33
Time Frame: Day 1 to Day 729
Population: as for outcome 33
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
participants
  PROTEIN, URINE, low: number analyzed (Participants) | 143 | 150
  PROTEIN, URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  PROTEIN, URINE, high: number analyzed (Participants) | 143 | 150
  PROTEIN, URINE, high | 0 | 0
  GLUCOSE, URINE, low: number analyzed (Participants) | 142 | 152
  GLUCOSE, URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  GLUCOSE, URINE, high: number analyzed (Participants) | 142 | 152
  GLUCOSE, URINE, high | 0 | 0
  BLOOD, URINE, low: number analyzed (Participants) | 147 | 154
  BLOOD, URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  BLOOD, URINE, high: number analyzed (Participants) | 147 | 154
  BLOOD, URINE, high | 0 | 0
  Red blood cells (RBC), URINE, low: number analyzed (Participants) | 152 | 156
  Red blood cells (RBC), URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  Red blood cells (RBC), URINE, high: number analyzed (Participants) | 152 | 156
  Red blood cells (RBC), URINE, high | 58 | 55
  White blood cells (WBC), URINE, low: number analyzed (Participants) | 152 | 156
  White blood cells (WBC), URINE, low | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value
  White blood cells (WBC), URINE, high: number analyzed (Participants) | 152 | 156
  White blood cells (WBC), URINE, high | 46 | 59

44. Secondary Outcome: Number of Participants With Other Marked Chemistry Laboratory Abnormalities in the Double Blind Period
Description: as for outcome 34
Time Frame: Day 1 to Day 729
Population: as for outcome 30
Measure: Number; unit: participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 153 | 160
participants
  GLUCOSE, SERUM, low: number analyzed (Participants) | 151 | 159
  GLUCOSE, SERUM, low | 15 | 24
  GLUCOSE, SERUM, high: number analyzed (Participants) | 151 | 159
  GLUCOSE, SERUM, high | 3 | 2
  GLUCOSE, FASTING SERUM, low: number analyzed (Participants) | 137 | 124
  GLUCOSE, FASTING SERUM, low | 3 | 1
  GLUCOSE, FASTING SERUM, high: number analyzed (Participants) | 137 | 124
  GLUCOSE, FASTING SERUM, high | 3 | 1
  PROTEIN, TOTAL, low | 10 | 7
  PROTEIN, TOTAL, high | 2 | 3
  ALBUMIN, low | 4 | 5
  ALBUMIN, high | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value | NA — Pre-specified marked lab abnormalities criteria do not include this low/high end value

45. Secondary Outcome: Number of Participants With Abatacept Induced Antibody Response Over Time in the Double-blind Period
Description: Participants who experienced a positive antibody response relative to baseline (ECL Assay)
Time Frame: Day 365, Day 729
Population: All treated participants in the immunogenicity analysis population for Year 1.
  Note: Study terminated, Year 2 data not collected
Measure: Number; unit: Participants
Arm/Group | Abatacept IV | Placebo IV
Number analyzed (Participants) | 202 | 203
Participants
  Day 365, overall: number analyzed (Participants) | 199 | 176
  Day 365, overall | 7 | 9
  Day 729, overall: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to 56 days post last dose (assessed up to May 2018, approximately 66 months)
Arm/Group | Abatacept IV | Placebo IV
All-Cause Mortality (participants affected / at risk) | 7/202 | 6/203
Serious Adverse Events (participants affected / at risk) | 62/202 | 58/203
Other Adverse Events (participants affected / at risk) | 164/202 | 179/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept IV (N=202) | Placebo IV (N=203)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Lupus myocarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Serositis (General disorders) | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Genital herpes (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 5 | 4
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 15 | 6
Pyelonephritis (Infections and infestations) | 0 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Salmonella bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 4
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 5
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 1
Lupus encephalitis (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Depression (Psychiatric disorders) | 1 | 0
Psychogenic seizure (Psychiatric disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 4 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 2 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept IV (N=202) | Placebo IV (N=203)
Anaemia (Blood and lymphatic system disorders) | 20 | 23
Abdominal pain upper (Gastrointestinal disorders) | 9 | 14
Diarrhoea (Gastrointestinal disorders) | 47 | 46
Nausea (Gastrointestinal disorders) | 13 | 17
Vomiting (Gastrointestinal disorders) | 12 | 7
Oedema peripheral (General disorders) | 15 | 13
Pyrexia (General disorders) | 9 | 13
Bronchitis (Infections and infestations) | 18 | 26
Conjunctivitis (Infections and infestations) | 14 | 15
Gastroenteritis (Infections and infestations) | 12 | 17
Herpes zoster (Infections and infestations) | 20 | 18
Influenza (Infections and infestations) | 11 | 9
Nasopharyngitis (Infections and infestations) | 40 | 44
Pharyngitis (Infections and infestations) | 20 | 24
Upper respiratory tract infection (Infections and infestations) | 43 | 42
Urinary tract infection (Infections and infestations) | 45 | 38
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 16
Dizziness (Nervous system disorders) | 12 | 5
Headache (Nervous system disorders) | 24 | 23
Insomnia (Psychiatric disorders) | 13 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 24
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 10
Rash (Skin and subcutaneous tissue disorders) | 11 | 20
Hypertension (Vascular disorders) | 7 | 12
Hypotension (Vascular disorders) | 5 | 13

LIMITATIONS AND CAVEATS:
Study terminated early after review of Year 1 data. Only Year 2/LTE data captured within blind was analyzed. Outcomes related to renal responses were not calculated due to lack of data caused by the early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.